CLINICAL TRIAL: NCT06918678
Title: Feasibility and Preliminary Efficacy of Remotely Delivered Tai Chi on Older Adults' 24-Hour Movement Behaviors: A Crossover Randomized Controlled Trial
Brief Title: Feasibility and Efficacy of A Remote Tai Chi Program in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Zan Gao, Professor and Department Head, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00017966
Record Dates: First submitted 2025-03-21; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Aging
Keywords: Physical activity; Tai Chi; Quality of life; Sedentary behaviors; Sleep; 24-hour Movement Behaviors; Fear of Falling; Psychosocial Beliefs of Physical Activity; Subjective Psychological Well-being; Cognitive Flexibility
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi intervention condition (Experimental): (1) the Tai Chi intervention condition followed by the Usual Care condition, or (2) the Usual Care condition followed by the TC intervention condition. Participants in the Tai Chi intervention condition were asked to attend a remotely delivered Tai Chi program, consisting of two 60-minute sessions each week. The Usual Care condition required participants to maintain their regular activities without Tai Chi and not to change their routine. Each condition lasted 12 weeks with a 2-week washout period separating the conditions to minimize carryover effects.
  Interventions: Device: Tai Chi intervention
- Usual Care condition (Active Comparator): The Usual Care condition required participants to maintain their regular activities without Tai Chi and not to change their routine.
  Interventions: Other: Usual care condiition

INTERVENTIONS:
Device: Tai Chi intervention — The Tai Chi program was delivered virtually via Zoom by a certified Tai Chi instructor for 12 weeks. Tai Chi forms employed in the class was adapted from an evident-based fall prevention program - Tai Ji Quan: Moving for Better Balance. This program is a research-based Tai Chi balance training regimen. The program composed of core adapted Tai Chi movements and various therapeutic movements as well as breathing exercises
  Arms: Tai Chi intervention condition
Other: Usual care condiition — In the usual care condition, the investigators requested that participants maintain their regular activities during their time in the usual care condition. The participants were encouraged to refrain from Tai Chi, but not prohibited from engaging in Tai Chi, in the usual care period.
  Arms: Usual Care condition

SUMMARY:
This project is designed to explore the feasibility and preliminary efficacy of a remote Tai Chi program on older adults' 24-hour movement behaviors (i.e., physical activity, sedentary behavior and sleep patterns).

DETAILED DESCRIPTION:
This study employed a 26-week cross-over, randomized control trial design in which each participant was assigned to one of two condition (i.e., 10 participants/cohort, 2 cohorts/condition) sequences at baseline: 1) the Tai Chi intervention condition then the usual care condition; or 2) usual care condition then intervention condition. The intervention condition requested participants participate in remote Tai Chi program for 60 minutes/session 2 times/week beyond their usual care. The usual care condition asked participants to maintain regular activities without Tai Chi and not to change their regular activity routine. Each condition lasted 12 weeks, with a 2-week washout separating treatments. The researchers monitored intervention fidelity via monthly follow-up phone calls.

ELIGIBILITY:
Eligible participants met the following inclusion criteria: 1) aged 60 years or older; 2) basic English communication skills; 3) without cognitive impairments or physical/mental dis-abilities that might limit their ability to practice TC, 4) computer/smartphone with internet access; and 5) provided informed consent. Participants who lacked the capacity to consent or had any medical condition that could make it potentially unsafe to be in an unsupervised physical space were excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility | Baseline, week 13, week 14, and week 26
  The investigators tracked participants' online attendance and let them complete a post-intervention satisfaction survey to assess acceptability and feasibility of the program. After the intervention, the investigators distributed a satisfaction survey including multiple choice questions and open-ended questions to the participants to evaluate their satisfaction and acceptability of the program.

SECONDARY OUTCOMES:
Physical activity | Baseline, week 12, week 14, and week 26
  Fitbit Inspire 3 Tracker owned by Google (Mountain View, California), a commercially available accelerometer-based activity tracker, was used to evaluate 24-hour movement behaviors. The participants received the device by mail, and the Fitbit tracker was given to the participants as an incentive to complete the study. The participants were encouraged to wear the Fitbit on their non-dominant wrist throughout the day, except for battery charging of the device, showering, and deep-water activities. The Inspire 3 tracked participants' physical activity (lightly active, fairly active, and very active).
Sedentary time | Baseline, week 12, week 14, and week 26
  Fitbit Inspire 3 Tracker owned by Google (Mountain View, California), a commercially available accelerometer-based activity tracker, was used to evaluate 24-hour movement behaviors. The participants received the device by mail, and the Fitbit tracker was given to the participants as an incentive to complete the study. The participants were encouraged to wear the Fitbit on their non-dominant wrist throughout the day, except for battery charging of the device, showering, and deep-water activities. The Inspire 3 tracked participants' sedentary time.
Sleep | Baseline, week 12, week 14, and week 26
  Fitbit Inspire 3 Tracker owned by Google (Mountain View, California), a commercially available accelerometer-based activity tracker, was used to evaluate 24-hour movement behaviors. The participants received the device by mail, and the Fitbit tracker was given to the participants as an incentive to complete the study. The participants were encouraged to wear the Fitbit on their non-dominant wrist throughout the day, except for battery charging of the device, showering, and deep-water activities. The Inspire 3 tracked participants' sleep.
Fear of Falling | Baseline, week 12, week 14, and week 26
  A shortened version of the Falls Efficacy Scale-International (Short FES-I) was used to assess fear of falling. This 7-item short FES-I has demonstrated excellent reliability (Cronbach's alpha 0.92) comparable to the original 16-item FES-I. The seven items evaluate the concerns of falling when carrying out daily activities such as getting dressed, taking a bath, or going out to a social event. Each item was rated on a 4-point Likert scale (1= "Not at all concerned" to 4= "Very concerned"). The total scores are summed from the questionnaire, and range from 7-28, with higher scores indicating more concerns about falling.
Older People's Quality of Life | Baseline, week 12, week 14, and week 26
  Quality of life was assessed by the brief Older People's Quality of Life questionnaire also known as the OPQOL-BRIEF. The OPQOL-BRIEF questionnaire has 13 items, with a preliminary single item on global quality of life. Each of the 13 items is scored Strongly agree=1, Agree=2, Neither=3, Disagree=4, Strongly disagree=5. The items are summed for a total OPQOL-Brief score, then positive items are reverse coded, so that higher scores represented higher quality of life.
Psychosocial Beliefs of Physical Activity | Baseline, week 12, week 14, and week 26
  Brief Psychosocial Scales [40] were used to assess psychosocial beliefs towards physical activity (PA). The four scales selected were: PA pros and cons (decisional balance, 8 items), PA self-efficacy (measuring confidence in PA, 6 items), PA social support (5 items), and PA enjoyment (4 items). All of these scales used a 5-point Likert format (1=not important, 5= extremely important). The PA decisional balance scale rates the importance of each statement to an individual's decision to be more active, with a higher score indicating more positive attitudes toward PA. A higher score on the PA self-efficacy, PA social support and PA enjoyments scales indicate more self-confidence, social support, and enjoyment during PA, respectively .
Cognitive Flexibility | Baseline, week 12, week 14, and week 26
  Card sorting, such as Wisconsin Card Sorting (WCS), has been often used to evaluate cognitive flexibility among older adults]. However, WCS takes approximately 30 minutes for older adults to complete, and it has been criticized for the potential stress it may cause older adults. Therefore, the investigators have adopted an online digital card sorting game (EFgo™), to assess participants' cognitive flexibility. The final score (ranging 0 -100, taking both trial accuracy and response time into account using a proprietary algorithm) of each participant was sent to the online database and retrieved by a research assistant for analysis.
Subjective Psychological Well-being | Baseline, week 12, week 14, and week 26
  Psychological wellbeing was assessed using the World Health Organization-Five Well-Being Index (WHO-5) scale remotely. The WHO-5 is a self-report instrument measuring mental well-being consisting of five statements relating to the past two weeks where each statement is rated on a 6-point scale, with higher scores indicating better mental well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided